CLINICAL TRIAL: NCT02560558
Title: Belatacept Immunosuppression Therapy in Post-Transplant Kidney Recipients: Comparison of 4-Week and 8-Week Dosing Intervals
Brief Title: Bela 8 Week Dosing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Idelberto Badell, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00082511
Record Dates: First submitted 2015-09-24; First posted 2015-09-25 (Estimated); Results first posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Kidney Transplantation
Keywords: Immunosuppression; Transplantation Immunology
MeSH Terms: interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Belatacept 8-weekly (Experimental): Subjects who are stable on belatacept therapy at least one year after a renal transplant will receive belatacept infusion intravenously (IV) at 5 mg/kg every 8 weeks.
  Interventions: Drug: Belatacept
- Belatacept 4-weekly (Active Comparator): Subjects who are stable on belatacept therapy at least one year after a renal transplant will receive belatacept infusion intravenously (IV) at 5 mg/kg every 4 weeks.
  Interventions: Drug: Belatacept

INTERVENTIONS:
Drug: Belatacept — Belatacept is an immunosuppressive medication and will be given as an intravenous infusion at a dose of 5 mg/kg at 4-weekly or 8-weekly intervals.
  Other Names: Nulojix

SUMMARY:
The purpose of this study is to transition patients who have been stable on Belatacept for one year after kidney transplant from standard 4-week to an investigational 8-week belatacept dosing schedule. The investigators hypothesize that renal function and acute rejection rates will be non-inferior with 8-week belatacept dosing.

DETAILED DESCRIPTION:
The current dosing protocol for patients who have undergone a kidney transplant requires that Belatacept be given as an infusion every 4 weeks. The investigator wants to assess if the patients who have been stable for one year after transplant can be safely transitioned to an 8-week Belatacept infusion schedule. Renal function and any episodes of acute rejection will be closely monitored.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥18 years currently),
* First-time renal transplant recipients of either living donor or deceased donor,

  1. who were initiated on belatacept at the time of transplant and
  2. are at least one year post-transplant and off CNI therapy for at least 6 months.
* Patients at low immunologic risk, defined as

  1. patients with a first transplant who have a PRA < 50 against class I and class II antigens,
  2. no DSA (donor-specific antibodies),
  3. who have not had more than one episode of rejection, and
  4. no episodes of rejection within the last 6 months prior to enrollment, and
  5. no rejection with a grade of IIB or above.

Exclusion Criteria:

* Not first renal transplant, or multi-organ transplant recipient
* History of greater than one episode of biopsy-proven acute rejection, or of rejection of Banff 97 grade IIB or greater, or rejection within the last 6 months.
* Pregnancy (women of childbearing potential must use adequate contraception during study)
* Unwilling to receive all belatacept infusions at the Emory Transplant Center
* Calculated Glomerular Filtration Rate (GFR) less than 35.
* Serum creatinine at enrollment over 30% higher than 3 months (±4 weeks) prior to randomization
* HbA1C greater than 8 at enrollment
* Recent history of significant proteinuria (protein/Cr ratio >1)
* Non-standard belatacept dosing (e.g. dose other than 5 mg belatacept/kg body weight)
* Cellcept dose less than 500 mg po bid.
* Prednisone dose greater than 5mg po qd within 3 months of randomization
* Patients not currently taking prednisone
* Active infection, or antibiotic or antiviral drug therapy within 1 month of randomization
* Evidence of Cytomegalovirus (CMV) viremia or clinical CMV infection within last 3 months.
* Polyomavirus BK PCR (polymerase chain reaction) load greater then 4.3 (copy number greater than 20,0000) within 3 months of randomization
* Known hepatitis B surface antigen-positive or PCR-positive for hepatitis B (testing not required)
* Known HIV (human immunodeficiency virus infection) (testing not required)
* Presence of donor specific antibody by Luminex single antigen assessment, or panel reactivity (PRA) above 50%.
* History of substance abuse or psychiatric disorder not compatible with study adherence and follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2015-09; Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Idelberto Badell, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory Clinic, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

REFERENCES:
- [Derived] Badell IR, Parsons RF, Karadkhele G, Cristea O, Mead S, Thomas S, Robertson JM, Kim GS, Hanfelt JJ, Pastan SO, Larsen CP. Every 2-month belatacept maintenance therapy in kidney transplant recipients greater than 1-year posttransplant: A randomized, noninferiority trial. Am J Transplant. 2021 Sep;21(9):3066-3076. doi: 10.1111/ajt.16538. Epub 2021 Mar 17. PMID 33583120

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Belatacept 8-weekly | Belatacept 4-weekly
Started | 84 | 82
Completed | 77 | 76
Not Completed | 7 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 0 | 4
Not completed — Protocol Violation | 3 | 0
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Population: Only included participants that received intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Belatacept 8-weekly | Belatacept 4-weekly | Total
Number analyzed (Participants) | 81 | 82 | 163
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (13) | 52 (12) | 51 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 19 | 46
  Male | 54 | 63 | 117
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 36 | 32 | 68
  Non African American | 45 | 50 | 95
Region of Enrollment [Number; unit: participants]
  United States | 81 | 82 | 163

OUTCOME MEASURES:

1. Primary Outcome: Mean Estimated Glomerular Filtration Rate (eGFR) at 12 Months From Baseline
Description: The mean estimated Glomerular Filtration Rate (eGFR) will be calculated according to the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation using serum creatinine measurements and the patient's age, gender, and race. An eGFR below 60 ml/min/1.73 m^2 indicates lower renal function.
Time Frame: 12 months from baseline
Measure: Mean (95% Confidence Interval); unit: ml/min/1.73m^2
Arm/Group | Belatacept 8-weekly | Belatacept 4-weekly
Number analyzed (Participants) | 77 | 76
ml/min/1.73m^2 | 72.13 [70.14 to 74.12] | 72.65 [70.64 to 74.65]

2. Secondary Outcome: Number of Participants With Transplant Rejection at 6 Months and 12 Months Post Baseline
Description: The number of occurrences of transplant rejection at 6 months and 12 months from baseline will be recorded.
Time Frame: 6 months post baseline, 12 months post baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Belatacept 8-weekly | Belatacept 4-weekly
Number analyzed (Participants) | 77 | 76
Participants
  6 months post baseline | 3 | 1
  12 months post baseline | 4 | 2

3. Secondary Outcome: Number of Subjects With Grade IIA and Lower Rejections at 6 Months and 12 Months Post Baseline
Description: The number of subjects with Grade IIA and lower severity of rejection on the Banff 97 diagnostic categories will be recorded. The severity of acute rejections will be graded based on histopathological findings; Grade IA= significant interstitial infiltration and moderate tubulitis; Grade IB= significant interstitial infiltration and severe tubulitis; Grade IIA= mild to moderate intimal arteritis; Grade IIB= severe intimal arteritis and Grade III= transmural arteritis and/or fibrinoid change and necrosis of cells.
Time Frame: 6 months post baseline, 12 months post baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Belatacept 8-weekly | Belatacept 4-weekly
Number analyzed (Participants) | 77 | 76
Participants
  6 months post baseline | 3 | 1
  12 months post baseline | 4 | 2

4. Secondary Outcome: Number of Subjects With Grade IIB and Higher Rejections at 6 Months and 12 Months Post Baseline
Description: The number of subjects with Grade IIB and higher severity of rejection on the Banff 97 diagnostic categories will be recorded. The severity of acute rejections will be graded based on histopathological findings; Grade IA= significant interstitial infiltration and moderate tubulitis; Grade IB= significant interstitial infiltration and severe tubulitis; Grade IIA= mild to moderate intimal arteritis; Grade IIB= severe intimal arteritis and Grade III= transmural arteritis and/or fibrinoid change and necrosis of cells.
Time Frame: 6 months post baseline, 12 months post baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Belatacept 8-weekly | Belatacept 4-weekly
Number analyzed (Participants) | 77 | 76
Participants
  6 months post baseline | 0 | 0
  12 months post baseline | 0 | 0

5. Secondary Outcome: Number of Deaths at 6 Months and 12 Months Post Baseline
Description: The total number of subject deaths at 12 months from baseline will be recorded.
Time Frame: 6 months post baseline, 12 months post baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Belatacept 8-weekly | Belatacept 4-weekly
Number analyzed (Participants) | 77 | 76
Participants
  6 months post baseline | 0 | 1
  12 months post baseline | 0 | 2

6. Secondary Outcome: Number of Subjects That Experienced Graft Loss at 6 Moths and 12 Months Post Baseline
Description: The total number of subjects who experienced death censored graft loss at 6 months and 12 months from baseline will be recorded.
Time Frame: 6 months post baseline, 12 months from baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Belatacept 8-weekly | Belatacept 4-weekly
Number analyzed (Participants) | 77 | 76
Participants
  6 months post baseline | 0 | 0
  12 months post baseline | 0 | 0

7. Secondary Outcome: Number of Subjects With Human Leukocyte Antigen Donor Specific Antibodies (HLA DSA) at 6 Months and 12 Months Post Baseline
Description: The number of subjects who have circulating human leukocyte antigen donor specific antibodies (HLA DSA) at 12 months from baseline will be recorded.
Time Frame: 6 moths post baseline, 12 months post baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Belatacept 8-weekly | Belatacept 4-weekly
Number analyzed (Participants) | 77 | 76
Participants
  6 months post baseline | 2 | 0
  12 months post baseline | 3 | 0

8. Secondary Outcome: Number of Clinic Visits
Description: The number of clinic visits by the subjects at the end of 12 months from baseline will be recorded.
Time Frame: At 12 months from baseline
Population: Resources/tools not available for recording/tracking the data required to reliably report the outcome.
Arm/Group | Belatacept 8-weekly | Belatacept 4-weekly
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Subjects Needing Hospitalizations
Description: The number of subjects who had hospitalizations at the end of 12 months from baseline will be recorded
Time Frame: At 12 months from baseline
Population: Resources/tools not available for recording/tracking the data required to reliably report the outcome.
Arm/Group | Belatacept 8-weekly | Belatacept 4-weekly
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Number of Subjects Needing Transplant Biopsies at 12 Months Post Baseline
Description: The number of subjects needing transplant biopsies at 12 months from baseline will be recorded.
Time Frame: 12 months post baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Belatacept 8-weekly | Belatacept 4-weekly
Number analyzed (Participants) | 77 | 76
Participants | 5 | 2

11. Secondary Outcome: Cost Analysis
Description: The mean total cost of infusions received by each subject and those associated with round trip travel to the Emory Transplant Center (ETC) will be estimated using the distance between the residential addresses of subjects and the ETC.
Time Frame: At 12 months from baseline
Population: Resources/tools not available for recording/tracking the data required to reliably report the outcome.
Arm/Group | Belatacept 8-weekly | Belatacept 4-weekly
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 12 months post baseline
Description: Adverse events were captured through active surveillance via open ended questions by the research coordinator at each study visit in accordance with the Common Terminology Criteria for Adverse Events (CTCAE)
Arm/Group | Belatacept 8-weekly | Belatacept 4-weekly
All-Cause Mortality (participants affected / at risk) | 0/77 | 2/76
Serious Adverse Events (participants affected / at risk) | 9/81 | 10/82
Other Adverse Events (participants affected / at risk) | 23/81 | 27/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belatacept 8-weekly (N=81) | Belatacept 4-weekly (N=82)
Infectious Severe Adverse Events (Infections and infestations) | 5 (6) | 6 (8)
Non Infectious severe Adverse Events (General disorders) | 4 (4) | 4 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belatacept 8-weekly (N=81) | Belatacept 4-weekly (N=82)
Infectious Adverse Events (Infections and infestations) | 19 (27) | 24 (30)
Non melanoma skin cancer (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1)
Other (General disorders) | 4 (5) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/58/NCT02560558/Prot_SAP_000.pdf